CLINICAL TRIAL: NCT05551416
Title: Research and Development of New Strategies for the Early Detection and Prevention of Gastric Cancer in the Spanish Population: EpiGASTRIC/EDGAR Project.
Brief Title: The EpiGASTRIC/EDGAR Project: New Strategies for the Early Detection and Prevention of Gastric Cancer
Status: Recruiting | Type: Observational
Sponsor: EDUARDO ALBENIZ (Other)
Collaborators: Institut d'Investigacions Biomèdiques August Pi i Sunyer (IDIBAPS), Spain (Unknown); Fundació Clínic per a la Recerca Biomèdica (FCRB), Spain (Unknown); Miguel Servet Foundation/Navarrabiomed, Spain (Unknown); Barcelona Clinic Hospital (HCB), Spain (Unknown); Navarre University Hospital (HUN), Spain (Unknown); Navarre Health Research Institute (IdiSNA), Spain (Unknown); Carlos III Health Institute (ISCIII), Spain (Unknown); Spanish Society of Digestive Endoscopy (SEED) Foundation (Unknown); Spanish Association of Gastroenterology (AEG) (Unknown)
Responsible Party: Sponsor-Investigator, EDUARDO ALBENIZ, MD, PhD, Fundacion Miguel Servet
Organization: Fundacion Miguel Servet (Other)
Other Study IDs: HCB/2021/0482-PI_2021/76
Record Dates: First submitted 2022-09-06; First posted 2022-09-22 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Gastric Neoplasms; Gastric Cancer; Gastric Lesion
Keywords: Gastric Cancer; Premalignant gastric lesions; Biomarkers; Prevalence; Endoscopy; Multiomics
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Nucleic acids and proteins will be obtained from the biological samples.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- EPIGASTRIC: Patients with GC.
  Interventions: Other: Identification of risk factors; Other: Identification of biomarkers; Other: Identification of gastric cancer hereditary predisposition
- EDGAR 1: Symptomatic patients subjected to a diagnostic gastroscopy to study the prevalence of premalignant gastric lesions.
  Interventions: Other: Identification of risk factors; Other: Characterization of premalignant gastric lesions; Other: Identification of biomarkers
- EDGAR 2: Patients with premalignant gastric lesions and early gastric neoplasias treated by endoscopy resection.
  Interventions: Other: Identification of risk factors; Other: Characterization of premalignant gastric lesions; Other: Identification of biomarkers
- Negative control: Patients from "EDGAR 1" without gastric pathology or familial history of this neoplasia.
  Interventions: Other: Identification of risk factors; Other: Identification of biomarkers

INTERVENTIONS:
Other: Identification of risk factors — Demographics, life habits and risk factors studies
Other: Characterization of premalignant gastric lesions — Identification and characterization of premalignant gastric lesions through high definition endoscopic study. Concordance between endoscopic and histological classifications
  Groups: EDGAR 1; EDGAR 2
Other: Identification of biomarkers — Multiomic studies
Other: Identification of gastric cancer hereditary predisposition — Genomic studies for the identification of individuals with hereditary GC predisposition
  Groups: EPIGASTRIC

SUMMARY:
This study is a multicenter, prospective cohort study, which are planned to enroll at least 600 patients who diagnosed the primary gastric cancer (GC); around 50 patients with premalignant gastric lesions (PGLs) and early gastric neoplasias (EGC) treated by endoscopy resection; and no less than 600 healthy normal cohort participants, for more than 18 months in the Spanish population. All participants who enrolled in this registry will be questioned by the life habits survey; and clinical data and biological samples of these participants were analyzed in order to look for new diagnostic tools.

The aim of this study is to evaluate clinical, endoscopic and molecular approaches to identify individuals with high-risk of GC. Thus, it would be allow the adoption of preventive measures to reduce mortality through early detection and/or the reduction of its incidence.

DETAILED DESCRIPTION:
Gastric cancer (GC) is the fifth most common and the third more deadly cancer in the world. In Spain, the incidence is 7.8 cases per 100,000 inhabitants, being twice as frequent in men as in women. During 2020, 7.577 new cases were diagnosed and approximately 5201 deaths occurred (Spanish association against cancer, AECC). Most cases are diagnosed in an advanced stage with a 5-year survival rate lower than 30%, which highlights the great importance of an early diagnosis.

Thus, this study aims to evaluate clinical, endoscopic and molecular approaches to identify individuals with high-risk of GC.

Methods: Coordinate and prospective project that considers the gender dimension of population-based study within a collaborative network. It includes different but interrelated cohorts:

1. "EDGAR 1": symptomatic patients undergoing a diagnostic gastroscopy to study the prevalence of PGLs;
2. "EDGAR 2": PGLs and EGC with indication for endoscopic resection;
3. "EPIGASTRIC": patients diagnosed with GC;
4. CONTROLS: patients without gastric pathology or a familial history of GC, obtained from the cohort EDGAR1.

Although GC diagnosis has been characterized by endoscopy, there has been a strong demand for low or non-invasive methods of GC detection. In this sense, clinical information and biological samples obtained by less invasive methods will be collected prospectively from the participating centers. State-of-the-art high-definition endoscopy and multiomic techniques will be used to perform:

* Clinical studies: Study the prevalence of GC and PGLs and genetic and environmental predisposing factors. Evaluation of high-definition endoscopy efficacy in the detection of PGLs and EGC. Concordance between endoscopic and histological classifications of PGLs. Estimate the risk of PGLs progression according to the follow-up of the lesions. Identification of GC-high-risk individuals, based on clinical data, familial factors, PGLs and a life habits survey.
* Translational studies: Identify and validate nucleic acids and proteins as new biomarkers of GC and PGLs in biological samples obtained by low or non-invasive methods and comparison with those obtained from histological samples and with the traditional markers used in GC diagnosis.

Given the multicenter nature of this project, standard operating procedures (SOPs) have also been established for the collection, processing, storage, and management of biological samples, so that it is carried out in the same way in all participating centers.

The data will be collected on the REDCap-AEG online platform, which can be accessed by researchers from each center through an identification code, respecting the current Organic Law on Data Protection. For patient registries, a specific database has been designed for each subproject (EDGAR 1, EDGAR 2 and EPIGASTRIC). This guarantees the quality of the data and allows its verification, as it defines, classifies and illustrates the different parameters to be assessed by the participating researchers. Finally, it allows the codification and anonymization of the data entered, which guarantees compliance with the data protection law of this study.

Statistical analysis: The SPSS program (IBM, NY) and/or the R software (https://www.r-project.org/) will be used. The differences between qualitative variables will be compared using Fisher's test. The quantitative variables will be analyzed using a non-parametric test (Mann-Whitney or Kruskall-Wallis for unpaired samples and Wilcoxon for paired samples). A "p" value <0.05 will be considered statistically significant. All the registered variables will be studied to determine their association with the diagnosis by means of univariate and multivariate logistic regression analysis. In addition, through an interaction study, we will evaluate whether there are risk factors associated with the presence/prognosis of lesions that differentially affect subgroups of patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years-old.
* EDGAR 1 cohort: symptomatic patients undergoing a diagnostic gastroscopy for a prevalence study of PGLs.
* EDGAR 2 cohort: PGLs and early GC with indication for endoscopic resection.
* EPIGASTRIC cohort: patients diagnosed with GC.
* CONTROL cohort: patients without gastric pathology or a familial history of GC, obtained from the EDGAR 1.

Exclusion Criteria:

* Refusal of the patient to participate in the study.
* Medical, psychological or legal inability of the patient to enter the study.
* EDGAR1: Previous diagnosis of PGLs, previous gastric surgery, contraindication for gastroscopy or taking biopsies.
* EDGAR 2: Contraindication for resection/biopsy.
* EPIGASTRIC: gastric neoplasm other than adenocarcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — In accordance with both ministerial and European guidelines on the assessment of the gender dimension in biomedical research, and given the differential incidence between both sexes in relation to gastric cancer, we will carry out differential analyzes by sex in all work packages. They will especially be carried out in biomarkers and risk factors studies, in order to understand the influence of sex in the early diagnosis of gastric cancer. We estimate that the collection of cases of gastric cancer will be double in males, although in the EDGAR 1 cohort that will study the prevalence of premalignant gastric lesions, we will try to obtain balanced data for both sexes.
Study Population: This cohort study is designed to enroll the Spanish population patients who are diagnosed gastric cancer; symptomatic patients subjected to a diagnostic gastroscopy who have or not premalignant gastric lesions and early gastric neoplasias susceptible to be treated by endoscopy resection; and healthy control participants by multicenter-prospective registry. Nevertheless, the study will be open to international participation.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
New strategies for gastric cancer (GC) early diagnosis | Up to 10 years
  Prediction of risk factors and identification of new strategies for an early diagnosis of GC.

SECONDARY OUTCOMES:
Prevalence of premalignant gastric lesions (PGLs) | Up to 5 years
  Determine the prevalence of PGLs in the EDGAR 1 cohort.
Endoscopic characterization of PGLs | Up to 5 years
  Identification and characterization of PGLs through high definition endoscopic study, testing the concordance between endoscopic and histological classifications.
Identification of GC hereditary predisposition by a customize multigene panel | Up to 5 years
  Define de most effective strategy for the identification of individuals with hereditary GC predisposition. In order to perform a clinical validation of the candidate genes identified by whole exome sequencing according to previous results of the research team (Herrera-Pariente, et al. IJMS 2021), a customize multigene panel has been designed including 25 potentially germline genetic variants associated to hereditary GC and 13 genes already associated with a higher risk of GC. This panel has been already tested, by the research group, ensuring its viability.
Identification of GC risk factors from clinical data and a lifestyle survey | Up to 5 years
  Based on the endoscopic classifications of the lesions found, the demographic data of the patient and their lifestyle and diet habits obtained through a specific questionnaire, risk factors involved in the development of CG will be identified through logistic regression. The identified risk factors will be used to create a predictive model.
Discover and validation of new biomarkers for early diagnosis of GC | Up to 5 years
  Multiomic data analysis of solid and liquid biopsies of the different cohorts in order to discover new molecules susceptible to be used as early diagnosis biomarkers. Validate them as screening test of GC.
Characterization of the microbiome: 16S rRNA studies | Up to 5 years
  The DNA extracted in the different cohorts is subjected to 16S rRNA gene-targeted sequencing to validate this microbial composition profile as a candidate for a noninvasive GC screening test.

CONTACTS AND LOCATIONS:
Locations (15):
- Spain (15):
  - Hospital Comarcal de Inca, Palma de Mallorca, Balearic Islands
  - Hospital de Llevant, Porto Cristo, Balearic Islands
  - Hospital General de Granollers, Granollers, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Hospital Santos Reyes, Aranda de Duero, Burgos
  - Hospital de Mérida, Mérida, Extremadura
  - Hospital Universitario de Ourense, Ourense, Galicia
  - Hospital Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Josep Trueta, Girona
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Herrera-Pariente C, Montori S, Llach J, Bofill A, Albeniz E, Moreira L. Biomarkers for Gastric Cancer Screening and Early Diagnosis. Biomedicines. 2021 Oct 12;9(10):1448. doi: 10.3390/biomedicines9101448. PMID 34680565
- [Background] Herrera-Pariente C, Capo-Garcia R, Diaz-Gay M, Carballal S, Munoz J, Llach J, Sanchez A, Bonjoch L, Arnau-Collell C, Soares de Lima Y, Golubicki M, Jung G, Lozano JJ, Castells A, Balaguer F, Bujanda L, Castellvi-Bel S, Moreira L. Identification of New Genes Involved in Germline Predisposition to Early-Onset Gastric Cancer. Int J Mol Sci. 2021 Jan 28;22(3):1310. doi: 10.3390/ijms22031310. PMID 33525650